CLINICAL TRIAL: NCT05109559
Title: A Phase 1/2 Study to Evaluate the Safety Reactogenicity and Immunogenicity of Ad26.COV2.S Administered as a Heterologous Booster Vaccination in Adults 18 Years of Age and Older Following Single- or Two-Dose Vaccination With an Inactivated COVID-19 Vaccine
Brief Title: Ad26.COV2.S as a Heterologous Booster in Adults After Single- or Two-Dose of Inactivated COVID-19 Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: National Vaccine Institute, Thailand (Other); International Vaccine Institute (Other); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC31518COV2012
Record Dates: First submitted 2021-11-03; First posted 2021-11-05 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; COVID-19; booster; Heterologous
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Ad26.COV2.S given at the interval ≥ 90 days after completing 2 doses of either Sinovac or Sinopharm (Experimental): Study Part A is a prospective, multi-center, Phase 2 study to assess a booster dose (3rd dose) of Ad26.COV2.S as an IM injection in the deltoid muscle in adults who have completed the two-dose homologous primary series of inactivated vaccine of Sinovac or Sinopharm, 21 to 35 days apart and who meet eligibility criteria.
  In study part A1, a total of 360 adult volunteers aged 18 years or older, will receive the full-dose (5x10^10 vp) of the study product, at later (90 days or more) time interval since the 2nd dose and followed from Visit 1 (V1) to Visit 7 (V7) at 336 days.
  Interventions: Biological: Full dose of Ad26.COV2. 5x10^10vp
- Ad26.COV2.S given at 45-75 days after completing 2 doses of either Sinovac or Sinopharm (Experimental): Study Part A is a prospective, multi-center, Phase 2 study to assess a booster dose (3rd dose) of Ad26.COV2.S as an IM injection in the deltoid muscle in adults who have completed the two-dose homologous primary series of inactivated vaccine of Sinovac or Sinopharm, 21 to 35 days apart and who meet eligibility criteria.
  In study part A2, a total of 110 adult volunteers aged 18 years or older, will receive the full-dose (5x10^10 vp) of the study product, at early (45-75 days) time interval since the 2nd dose and followed from Visit 1 (V1) to Visit 7 (V7) at 336 days.
  Interventions: Biological: Full dose of Ad26.COV2. 5x10^10vp
- Half dose of Ad26.COV2.S given ≥ 90 days after completing 2 doses of either Sinovac or Sinopharm (Experimental): Study Part A is a prospective, multi-center, Phase 2 study to assess a booster dose (3rd dose) of Ad26.COV2.S as an IM injection in the deltoid muscle in adults who have completed the two-dose homologous primary series of inactivated vaccine of Sinovac or Sinopharm, 21 to 35 days apart and who meet eligibility criteria.
  In study part A3, a total of 110 adult volunteers aged 18 years or older, will receive the half-dose (2.5x10^10 vp) of the study product, at later (90 days or more) time interval since the 2nd dose and followed from Visit 1 (V1) to Visit 7 (V7) at 336 days.
  Interventions: Biological: Half dose of Ad26.COV2. 2.5x10^10vp
- Ad26.COV2.S given 28 days after receiving 1 dose of either Sinovac or Sinopharm (Experimental): Study Part B is a prospective, multi-center, open-label Phase 1/2 heterologous prime-boost study to assess the Ad26.COV2.S (full dose 5x10^10 vp) as the 2nd vaccination in subjects who are documented to all have received the 1st dose of Sinovac or all received the 1st dose of Sinopharm COVID-19 vaccine, with an interval of 28 days +/- 3 days, followed from Visit 1 (V1) to Visit 7 (V7) at 336 days.
  Interventions: Biological: Full dose of Ad26.COV2. 5x10^10vp

INTERVENTIONS:
Biological: Full dose of Ad26.COV2. 5x10^10vp — A booster dose (3rd dose) of Ad26.COV2.S as an IM injection in the deltoid muscle in adults.
  Arms: Ad26.COV2.S given at 45-75 days after completing 2 doses of either Sinovac or Sinopharm; Ad26.COV2.S given at the interval ≥ 90 days after completing 2 doses of either Sinovac or Sinopharm
Biological: Half dose of Ad26.COV2. 2.5x10^10vp — A booster dose (3rd dose) of Ad26.COV2.S as an IM injection in the deltoid muscle in adults.
  Arms: Half dose of Ad26.COV2.S given ≥ 90 days after completing 2 doses of either Sinovac or Sinopharm
Biological: Full dose of Ad26.COV2. 5x10^10vp — A booster dose (2nd dose) of Ad26.COV2.S as an IM injection in the deltoid muscle in adults.
  Arms: Ad26.COV2.S given 28 days after receiving 1 dose of either Sinovac or Sinopharm

SUMMARY:
This study aims to address evidence gaps regarding the safety, reactogenicity and immune responses of a heterologous boost of a single dose of Ad26.COV2.S (half or full dose) at pre-specified time intervals in recipients who are documented to have received either 1-dose or 2-doses (primary series completion) of inactivated COVID-19 vaccines, Sinovac and/or Sinopharm.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observer-blind Phase 1/2 adaptive study to assess the safety, reactogenicity, and immunogenicity of a booster dose of Ad26.COV2.S in adults ≥ 18 years of age in Study Part A and Part B. A total of 690 participants will be recruited. If the optional Group (A4) is feasible and enrolled, the total recruitment will be 800 participants. Priority enrolment is given to Groups A1 and A2, followed by Groups A3 and B1. Enrolment of groups are open-label allocation and assessor-masked.

The Study is divided into 2 Parts: Part A and B.

Study Part A is a prospective, multi-center, assessor-masked Phase 1/2 study to assess a booster dose (3rd dose) of Ad26.COV2.S as an IM injection in the deltoid muscle in adults who have completed the two-dose homologous primary series of inactivated vaccine of Sinovac or Sinopharm, 21 to 35 days apart and who meet eligibility criteria. Participants will receive either the full-dose (5x10^10 vp) or half-dose (2.5x10^10 vp) of the study product, and at early (45-75 days) or later (90-240 days) time interval and followed from Visit 1 (V1) to Visit 7 (V7) at 336 days.

A total of 580 adult volunteers aged 18 years or older, who have verified vaccination cards with documented completion of homologous primary vaccination series with either two doses of Adsorbed COVID-19 (inactivated) Sinovac (SV) or Sinopharm (SP) vaccine, against original and novel variants of SARS-CoV-2 will be enrolled. A 20% dropout rate is assumed. Enrolment is increased to 360 (300+20% dropout) for the safety assessment, to detect common adverse events with an event rate of 1%.

Part B is a prospective, multi-center, open-label, assessor-masked Phase 1/2 heterologous prime-boost study to assess the Ad26.COV2.S (full dose) as the 2nd vaccination in subjects who are documented to all have received the 1st dose of Sinovac or all received the 1st dose of Sinopharm COVID-19 vaccine, with an interval of 28 days or more, followed from Visit 1 (V1) to Visit 7 (V7) at 336 days.

Together with the Sponsor, the PIs will decide on the feasibility of enrolment of participants who all have already received 1 dose of Sinopharm or who all have received 1dose of Sinovac, based on current public health policy and vaccine coverage.

For safety assessment:

Adverse events (AEs) will be systematically collected at all clinic visits. Solicited AEs will be assessed in all subjects immediately (30 minutes) after each injection. Subjects (or with necessary supports) will record solicited AEs daily in the Diary Card for the seven days following injection. If a solicited AE is ongoing at a 7-day post-injection follow-up visit (Visit 2), or occurs after 7 days post-injection, the event will be recorded as AE and continued to be followed as per AE monitoring requirements.

Adverse events and special reporting situations, whether serious or non-serious, that are related to study procedures or that are related to non-investigational sponsor products will be reported from the time a signed and dated informed consent form (ICF) is obtained until the end of the study/early withdrawal. All other unsolicited AEs will be reported from the time of vaccination until completion of the participant's last study-related procedure. All AESIs, SAEs, and AEs leading to discontinuation from the study (regardless of the causal relationship) are to be reported from the moment of vaccination until completion of the participant's last study related procedure.

For immunological assessment:

Primary objectives

1. To assess the IgG immune response against the Spike protein of SARS-CoV-2, measured by ELISA and compared with baseline (pre-boost titer) at Days 28, 84, 168 and 336 following either half dose (2.5x10^10 virus particles (vp)) or full dose (5x10^10 vp) of Ad26.COV2.S vaccination at pre-specified time intervals in adults who have already received either one-dose or two-doses of an inactivated COVID-19 vaccine.
2. To assess a subset for functional (neutralizing) humoral immune responses elicited by each of the regimens as measured by pseudovirus neutralization assay, IgG at baseline, Days 28, 84, 168 and 336 following Ad26.COV2.S vaccination.

Secondary objective

1. To assess a subset for functional (neutralizing) humoral immune responses elicited by each of the regimens as measured by microneutralization neutralization assay, IgG at baseline, Days 28, 84, 168 and 336 following Ad26.COV2.S vaccination.

Exploratory Objectives

1. To characterize PCR-confirmed COVID-19 breakthrough infections following booster vaccination by assessing anti-S and anti-N IgG.
2. To characterize cellular immune responses including Th1/Th2.
3. To consider statistical tests of noninferiority in comparing the different study arms.
4. To assess Adenovirus 26 neutralizing antibodies at baseline if feasible.

Study duration: Subjects will be followed for approximately 336 days following Ad26.COV2.S vaccination. The total study period will be 18 months, including 12-month follow-up period.

The Clinical Data Management System, including eCRFs, statistical analysis and data archival are under the responsibility of the center of excellence for Biomedical and Public Health Informatics (BIOPHICS), the center of data management for clinical research at the Faculty of Tropical Medicine, Mahidol University.

Based on the final protocol of the study, a comprehensive set of CRFs/eCRFs will be prepared to capture all the relevant data required for analysis and reporting.

Information about COVID-19 disease, correlates of immunity, safety, and local epidemiology and public health context regarding the new SARS-CoV-2 virus are rapidly evolving during the pandemic. Therefore, it is critical to recognize that the approach outlined in this document may be adapted as new data, expert consensus and public health policies evolve.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must meet all inclusion criteria to be enrolled and participate in the study, as follows:

1. Adult male or female aged 18 years or more on the day of signing the ICF, confirmed by identification cards.
2. Verified, documentation of past COVID-19 vaccination i. Study Part A: having completed the 2-dose homologous primary regimen (21 to 35 days apart) of inactivated COVID-19 vaccine of either Sinovac-Sinovac OR Sinopharm-Sinopharm ii. Study Part B: having received one dose of inactivated COVID-19 vaccine of either Sinovac or Sinopharm with the appropriate interval period
3. Women of childbearing potential who are test negative with a highly sensitive urine pregnancy test at Visit 1, prior to study vaccine administration.
4. Subject has provided written informed consent prior to performance of any study-specific procedures and is willing and has means to be contacted and to contact the investigator during the study.
5. In the investigator's clinical judgment, the participant is in good health, or has stable and well-controlled medical conditions.
6. Participant agrees to not donate bone marrow, blood, and blood products from the study vaccine administration until 3 months after receiving the study vaccine.

Exclusion Criteria:

Potential participants who meet any of the following exclusion criteria will be excluded from enrolment and participation in the study:

1. The participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection), or is a patient under investigation (PUI) or has a body temperature ≥38.0ºC (100.4°F) within 24 hours prior to the planned study vaccination. Assignment may be made at a later date is permitted at the discretion of the investigator. Please notify the Sponsor (or medical monitor) of this decision.
2. Contraindication to Ad26.COV2.S according to labelling of the product. For example, if the participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine;refer to the IB (IB Edition 5 Ad26.COV2.S 2021 and its addenda).
3. Pregnant or planning to become pregnant within 3 months after study vaccine administration
4. Participant has a history or current condition as follows

   1. Known documented history of COVID-19 infection prior to enrollment
   2. Any confirmed or suspected immunosuppressive or immunodeficient state.
   3. Heparin-induced thrombocytopenia or thrombosis in combination with thrombocytopenia.
   4. Acute polyneuropathy (e.g. Guillain-Barré syndrome).
   5. Capillary leak syndrome
   6. Contraindication to IM injections and blood draws e.g., bleeding disorders.
   7. An underlying clinically significant acute or chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well being) or that could prevent, limit, or confound the protocol-specified assessments.
   8. Major psychiatric illness which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures.
5. If the participant received or plans to receive:

   1. Licensed live attenuated vaccines - within 28 days before or after planned administration of study vaccine.
   2. Other licensed (not live) vaccines - within 14 days before or after planned administration of study vaccine.
   3. Treatment with immunoglobulins (Ig) in the 3 months or exogenous blood products (autologous blood transfusions are not exclusionary) in the 4 months before the planned administration of the study vaccine or has any plans to receive such treatment during the study.
6. If the participant cannot communicate reliably with the investigator, or, in the opinion of the investigator, is unlikely to adhere to the requirements of the study or is unlikely to complete the full course of vaccination and observation.
7. Employee of the study center directly involved with the proposed study or with study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited reportable local adverse event after vaccination | Day 0 through Day 7
  Frequency and percentage of solicited reportable local adverse events (pain or tenderness, erythema, swelling or induration) of vaccination
Frequency of solicited reportable systemic adverse event after vaccination | Day 0 through Day 7
  Frequency and percentage of solicited reportable systemic adverse events (fever, headache, fatigue or malaise, myalgia, arthralgia, nausea or vomitting) of vaccination
Frequency of all unsolicited AEs | : Day 0 through Day 336
  Frequency and percentage of all unsolicited AEs
GMT Anti-S IgG at baseline | Day 0
  GMT Anti-S IgG at baseline
GMT Anti-S IgG at 7 days after vaccination in subset subjects | Day 7
  GMT Anti-S IgG at 7 days after vaccination in subset subjects
GMT Anti-S IgG at 14 days after vaccination in subject subjects | Day 14
  GMT Anti-S IgG at 14 days after vaccination in subset subjects
GMT Anti-S IgG at 28 days after vaccination | Day 28
  GMT Anti-S IgG at 28 days after vaccination
GMT Anti-S IgG at 84 days after vaccination | Day 84
  GMT Anti-S IgG at 84 days after vaccination
GMT Anti-S IgG at 168 days after vaccination | Day 168
  GMT Anti-S IgG at 168 days after vaccination
GMT Anti-S IgG at 336 days after vaccination | Day 336
  GMT Anti-S IgG at 336 days after vaccination
GMFR changed from baseline in anti-S IgG GMT at 28 days after vaccination | Day 28
  GMFR changed from baseline in anti-S IgG GMT at 28 days vaccination
GMFR changed from baseline in anti-S IgG GMT at 84 days after vaccination | Day 84
  GMFR changed from baseline in anti-S IgG GMT at 84 days vaccination
GMFR changed from baseline in anti-S IgG GMT at 168 days after vaccination | Day 168
  GMFR changed from baseline in anti-S IgG GMT at 168 days vaccination
GMFR changed from baseline in anti-S IgG GMT at 336 days after vaccination | Day 336
  GMFR changed from baseline in anti-S IgG GMT at 336 days vaccination
Anti-S IgG Seroresponses changed from baseline at 28 days after vaccination | Day 28
  Frequency and percentage of participants with seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline at 28 days after vaccination
Anti-S IgG Seroresponses changed from baseline at 84 days after vaccination | Day 84
  Frequency and percentage of participants with seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline at 84 days after vaccination
Anti-S IgG Seroresponses changed from baseline at 168 days after vaccination | Day 168
  Frequency and percentage of participants with seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline at 168 days after vaccination
Anti-S IgG Seroresponses changed from baseline at 336 days after vaccination | Day 336
  Frequency and percentage of participants with seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline at 336 days after vaccination

SECONDARY OUTCOMES:
GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at baseline | Day 0
  GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at baseline
GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 28 days after Ad26.COV2.S vaccination | Day 28
  GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 28 days after Ad26.COV2.S vaccination
GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 84 days after Ad26.COV2.S vaccination | Day 84
  GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 84 days after Ad26.COV2.S vaccination
GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 168 days after Ad26.COV2.S vaccination | Day 168
  GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 168 days after Ad26.COV2.S vaccination
GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 336 days after Ad26.COV2.S vaccination | Day 336
  GMT measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) Neutralizing antibody titer 50 at 336 days after Ad26.COV2.S vaccination
GMFR changed from baseline (pre-boost titer) in NT50 measured by pNA and mNA against SARS-CoV-2 Delta and Wildtype at 28 days after Ad26.COV2.S vaccination | Day 28
  GMFR changed from baseline (pre-boost titer) in NT50 measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) against SARS-CoV-2 Delta and Wildtype) at 28 days after Ad26.COV2.S vaccination among those positives by pNA assay
GMFR changed from baseline (pre-boost titer) in NT50 measured by pNA and mNA against SARS-CoV-2 Delta and Wildtype at 84 days after Ad26.COV2.S vaccination | Day 84
  GMFR changed from baseline (pre-boost titer) in NT50 measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) against SARS-CoV-2 Delta and Wildtype) at 84 days after Ad26.COV2.S vaccination among those positives by pNA assay
GMFR changed from baseline (pre-boost titer) in NT50 measured by pNA and mNA against SARS-CoV-2 Delta and Wildtype at 28 days after Ad26.COV2.S vaccination | Day 168
  GMFR changed from baseline (pre-boost titer) in NT50 measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) against SARS-CoV-2 Delta and Wildtype) at 168 days after Ad26.COV2.S vaccination among those positives by pNA assay
GMFR changed from baseline (pre-boost titer) in NT50 measured by pNA and mNA against SARS-CoV-2 Delta and Wildtype at 28 days after Ad26.COV2.S vaccination | Day 336
  GMFR changed from baseline (pre-boost titer) in NT50 measured by pseudovirus neutralization assay (pNA) and microneutralization assay (mNA) against SARS-CoV-2 Delta and Wildtype) at 336 days after Ad26.COV2.S vaccination among those positives by pNA assay

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, MD, Study Chair — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, 420/6 Ratchawithi Road, Ratchathewi,, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muangnoicharoen S, Wiangcharoen R, Lawpoolsri S, Nanthapisal S, Jongkaewwattana A, Duangdee C, Kamolratanakul S, Luvira V, Thanthamnu N, Chantratita N, Thitithanyanont A, Anh Wartel T, Excler JL, Ryser MF, Leong C, Mak TK, Pitisuttithum P. Heterologous Ad26.COV2.S booster after primary BBIBP-CorV vaccination against SARS-CoV-2 infection: 1-year follow-up of a phase 1/2 open-label trial. Vaccine. 2024 Jul 25;42(19):3999-4010. doi: 10.1016/j.vaccine.2024.05.010. Epub 2024 May 13. PMID 38744598
- [Derived] Muangnoicharoen S, Wiangcharoen R, Nanthapisal S, Kamolratakul S, Lawpoolsri S, Jongkaewwattana A, Thitithanyanont A, Luvira V, Chinwangso P, Thanthamnu N, Chantratita N, Lim JK, Anh Wartel T, Excler JL, Ryser MF, Leong C, Mak TK, Pitisuttithum P. Single Ad26.COV2.S booster dose following two doses of BBIBP-CorV vaccine against SARS-CoV-2 infection in adults: Day 28 results of a phase 1/2 open-label trial. Vaccine. 2023 Jul 19;41(32):4648-4657. doi: 10.1016/j.vaccine.2023.06.043. Epub 2023 Jun 15. PMID 37344265